CLINICAL TRIAL: NCT00235092
Title: A Prospective, Randomized, Multi-Center Comparison of the Cypher Sirolimus-Eluting and the Taxus Paclitaxel-Eluting Stent Systems.
Brief Title: The REALITY Study - Head-to-Head Comparison Between Cypher and Taxus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC03-02
Record Dates: First submitted 2005-10-04; First posted 2005-10-10 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cypher Sirolimus-Eluting Stent
Device: Taxus Paclitaxel-Eluting Stent

SUMMARY:
The main objective of this study is to compare the performance of the Cypher sirolimus-eluting and the Taxus paclitaxel-eluting stent systems in a prospective, multi-center, randomized clinical study.

DETAILED DESCRIPTION:
This is a prospective, randomized study conducted at 90 centers in Europe, Latin-America and Asia. A total of 1335 patients will be entered into the study and will be randomized on a 1:1 basis to either the sirolimus-eluting or the paclitaxel-eluting stent system. All patients will have repeat angiography at eight months and will be followed for 24 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
2. Treatment of up to two de novo native coronary artery lesions in a maximum of two major coronary arteries;
3. Ostial lesions;
4. Bifurcations;
5. Target vessel diameter of both lesions must be >=2.25mm and <=3.0mm in diameter (visual estimate);
6. One target lesion must be at least 15 mm in length and the second lesion has to be at least 10 mm in length with no upper limit on either;
7. Target lesion stenosis for both lesions is >50% and <100% (visual estimate).

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 72 hours and the CK and CK-MB enzymes remain above normal at the time of treatment;
2. Has unstable angina classified as Braunwald A I-II-III;
3. Any of the lesions is an unprotected left main coronary disease with >=50% stenosis;
4. Angiographic evidence of thrombus within target lesion;
5. Heavily calcified lesion and/or calcified lesion, which cannot be successfully predilated (applies to both lesions);
6. Documented left ventricular ejection fraction <=25%;

8. Totally occluded vessel (TIMI 0 level) (applies to both lesions);

9. Prior stent within 10mm of target lesion (applies to both lesions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1335
Dates: Start 2003-08; Study Completion 2006-03

PRIMARY OUTCOMES:
The primary endpoint of the study is angiographic in-lesion binary restenosis rate at 8 months follow-up as determined by QCA.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Morice, MD, Principal Investigator — Institut Hospitalier Jacques Cartier
Locations (1):
- Institut Hospitalier Jacques Cartier, Massy, France

REFERENCES:
- [Result] Morice MC, Colombo A, Meier B, Serruys P, Tamburino C, Guagliumi G, Sousa E, Stoll HP; REALITY Trial Investigators. Sirolimus- vs paclitaxel-eluting stents in de novo coronary artery lesions: the REALITY trial: a randomized controlled trial. JAMA. 2006 Feb 22;295(8):895-904. doi: 10.1001/jama.295.8.895. PMID 16493102